CLINICAL TRIAL: NCT03955419
Title: Randomized Controlled Trial Comparing Preoperative Oral Carbohydrate Loading With Standard Overnight Fasting in Gynecologic Surgery.
Brief Title: Preoperative Oral Carbohydrate Loading in Gynecologic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunah Cho, MD (Other)
Responsible Party: Sponsor-Investigator, Eunah Cho, MD, Clinical Assistant Professor, Kangbuk Samsung Hospital
Organization: Kangbuk Samsung Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KBSMC 2019-04-015-001
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Postoperative Recovery
MeSH Terms: interventions — Long-Term Synaptic Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Participants in the control group will be fasted from midnight until surgery.
- Study group (Experimental): Participants will receive 800 mL of carbohydrate beverage (12.8% carbohydrates, 50 kcal/100 mL, 290 mOsm/kg). They will drink this beverage freely, starting from the evening before surgery until 2 hours before surgery.
  Interventions: Dietary Supplement: NO-NPO (Daesang WelLife Co., Ltd., Korea)

INTERVENTIONS:
Dietary Supplement: NO-NPO (Daesang WelLife Co., Ltd., Korea) — 800 mL of carbohydrate beverage consists of 12.8% carbohydrates, 50 kcal/100 mL, 290 mOsm/kg.
  Arms: Study group

SUMMARY:
The advantage of carbohydrate loading in minimally invasive surgeries are not well established. We designed this study to evaluate whether preoperative oral carbohydrate improve postoperative recovery after laparoscopic gynecologic surgeries.

DETAILED DESCRIPTION:
This study will be conducted in the female adult patient scheduled for laparoscopic gynecologic surgery for benign or premalignant condition. Patients with American Society of Anesthesiologist physical status classification I-II, not pregnant or on lactation will be included. Patients with underlying disease that will delay gastric emptying (GERD, history of gastrointestinal surgery, diabetes), or contraindicated to NSAID or opioid, psychiatric or mental disorders, alcoholism, or drug abuse will be excluded.

Participants will be randomized into 2 group: the control group and the study group. Randomization will be conducted via random block with stratification generated by the http://www.randomization.com with 1:1 allocation. The sequence will be kept in opaque, sealed envelopes until the day before the study date. One investigator, not involved in the outcome assessment, opened the envelope on the day before the surgery, and allocated participants in each group.

After having regular diet until the evening before surgery, participants allocate in the control group were kept fasted from midnight until surgery. Participants in the study group will receive 800 mL of carbohydrate beverage (12.8% carbohydrates, 50 kcal/100 mL, 290 mOsm/kg). The participants in the study group will freely drink carbohydrate beverage starting from the evening before surgery up to 2 hours before surgery.

The postoperative quality of recovery (QoR) score, time to readiness to discharge, patient satisfaction, postoperative nausea and vomiting, change in body weight, and insulin resistance will be assessed.

ELIGIBILITY:
Inclusion Criteria:

age between 18 and 70 years American Society of Anesthesiologists physical status (ASAPS) classification I-II absence of pregnancy or lactation at the time of surgery.

Exclusion Criteria:

suspicious delayed gastric emptying such as GERD or gastrointestinal surgery metabolic disorders such as diabetes known contraindications to NSAID or opioid physically disabled severe psychiatric or mental disorders alcoholism, drug abuse

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with indication for laparoscopic gynecologic surgery for benign or premalignant gynecologic conditions
Enrollment: 88 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Quality of recovery (QoR)-15 score | 2 days after surgery
  This score measures the quality of recovery after surgery in 2 dimensions, which are the physical well-being (in 9 items) and mental well-being (6 items). Each item is rated from 0 (poor) to 10 (excellent). A sum of each score represents the QoR of the patients.

SECONDARY OUTCOMES:
time to readiness to discharge (TRD) | 2 days after surgery
  This measures the time when the patients are ready to discharge from the hospital after surgery. It assesses five criteria: (1) tolerance of oral intake, (2) recovery of lower gastrointestinal function, (3) adequate pain control with oral analgesia, (4) ability to mobilize and perform self-care, and (5) clinical examination and laboratory tests. TRD is defined by the time from the operation end time to the time when time to readiness to discharge criteria is fulfilled.

CONTACTS AND LOCATIONS:
Overall Officials: Eunah Cho, M.Dm., Principal Investigator — Kangbuk Samsung Hospital
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cho EA, Lee NH, Ahn JH, Choi WJ, Byun JH, Song T. Preoperative Oral Carbohydrate Loading in Laparoscopic Gynecologic Surgery: A Randomized Controlled Trial. J Minim Invasive Gynecol. 2021 May;28(5):1086-1094.e1. doi: 10.1016/j.jmig.2020.12.002. Epub 2020 Dec 10. PMID 33310170